CLINICAL TRIAL: NCT04291378
Title: The DBCG Proton Trial. Adjuvant Breast Proton Radiation Therapy for Early Breast Cancer Patients: The Skagen Trial 2, a Clinically Controlled Randomised Phase III Trial
Brief Title: The DBCG Proton Trial: Photon Versus Proton Radiation Therapy for Early Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Breast Cancer Cooperative Group (Other)
Responsible Party: Principal Investigator, Birgitte Offersen, Professor, phd, Danish Breast Cancer Cooperative Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DBCG Proton trial
Record Dates: First submitted 2020-02-24; First posted 2020-03-02 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Early Breast Cancer; Radiation Associated Cardiac Failure
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients are randomised between 2 arms with different types of radiation therapy, and patients in both arms have similar follow up
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Photon radiation therapy (Active Comparator): The patient is treated with standard radiation therapy based on photons
  Interventions: Radiation: Proton versus photon radiation therapy
- Proton radiation therapy (Experimental): The patient is treated with experimental radiation therapy based on protons
  Interventions: Radiation: Proton versus photon radiation therapy

INTERVENTIONS:
Radiation: Proton versus photon radiation therapy — The intervention is proton radiation therapy versus photon radiation therapy

SUMMARY:
The majority of early breast cancer patients are treated with adjuvant radiation therapy (RT) as part of their multimodal therapy. The aim of the RT is to lower the risk of local, regional and distant failure and improve survival. Modern RT is been provided with photon therapy. Now, more proton therapy facilities are opened, including in Denmark. Proton RT may have the potential to cause lower dose to heart and lung during breast RT. This trial will randomise patients between standard photon RT versus experimental proton RT. The primary endpoint is 10 year risk of heart disease.

DETAILED DESCRIPTION:
Adjuvant breast cancer radiation therapy (RT) is standard for all patients operated with breast conservation and for patients diagnosed with large tumours and/or node-positive disease. Around 65% of all breast cancer patients treated with RT have whole breast RT without nodal RT, whilst the remaining 35% are treated with loco-regional RT (target is breast / chest wall and regional nodal volumes). RT leads to fewer local and regional recurrences, a decrease in breast cancer death and improves overall survival. Since 2014, when the DBCG IMN study showed overall survival gain from internal mammary node (IMN) RT, IMN RT has been standard for all high-risk patients in Denmark. IMN RT causes a significant increase in dose to the heart and lung, thus heart and lung sparing RT techniques based on deep inspiration breath hold (DIBH), volumetric arc therapy and tomotherapy are increasingly used to lower dose to heart and lung whilst maintaining dose to breast and nodal targets. These advanced techniques are used in all DBCG departments routinely. Despite using advanced RT techniques, some patients still receive high RT dose to heart and lung.

Proton therapy (PT) has not been widely used nor investigated for adjuvant breast cancer RT, because there are only few proton centres. However, due to the properties of PT it is possible to achieve optimal dose coverage of relevant targets and at the same time ensure low dose to organs at risk compared with photon RT. In an energy-dependent manner, PT will deposit the majority of its dose in tissue depths defined by the Bragg peak. In practice, this translates into i) the ability to deliver the peak energy to target volumes of irregular 3-dimensional shape using pencil-beam scanning technology, ii) a sharp dose fall-off following deposition of energy in the target and iii) reduction of the integral dose to the patient. Within millimeters, the exit dose drops off from 90% to 10%, resulting in the virtual absence of an exit dose. The effectiveness, safety and feasibility of PT has been reported in few small cohort studies with limited follow up, and there is a lack of clinically controlled randomised trials documenting benefit from PT, evaluated either as higher tumour control and/or as fewer morbidities.

This trial tests standard photon RT versus experimental proton RT for selected early breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient operated for early breast cancer with indication for radiation therapy, where standard planning shows a mean heart dose 4 Gy or more and/or a V20 lung of 37% or more.
* Boost (breast, chest wall and nodal), breast reconstruction (any type, except implants with metal), connective tissue disease, post-operative surgical complications, any breast size and seromas are allowed
* Patient with previous non-breast malignancy is accepted if the patient has been without disease minimum 5 years, and the treating oncologist estimates a low risk of recurrence.
* Life expectancy minimum 10 years

Exclusion Criteria:

* previous breast cancer/ductal carcinoma in situ,
* Previous RT to the chest region
* Pregnant or lactating
* Conditions indicating that the patient cannot go through the RT or follow up
* Patients with Pacemaker or defibrillator are excluded until a guideline for handling them has been developed at the DCPT
* Unknown non-tissue implants upstream of the target volume. NB. all such non-tissue, non-metal objects must be delivered to the DCPT for stopping power determination and evaluation at least a week prior to radiation start.
* Metal implants in the radiation area, including metal in implants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1502 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2037-06-01 (Estimated)

PRIMARY OUTCOMES:
Radiation associated ischaemic and valvular heart disease | 10 years after RT
  The following incidences heart diseases according to ICD10: ischaemic heart disease codes I20-25 and valvular heart disease codes I00-09, I01.0, I09.2, I34-39

SECONDARY OUTCOMES:
Radiation associated second cancer | 10 years after RT
  Incidences of second cancer associated with the RT: lung, esophagus, thyroid, sarcoma, contralateral breast
Distant failure | 10 years after RT
  Incidences of distant failures, i.e. cancer recurrence outside the loco-regional region
Acute radiation associated morbidity | within 6 months after RT
  According to CTC version 4.0: Incidences of radiation dermatitis, itching, pain, fatigue, dyspnea, cough, pneumonitis, dysphagia, increased sensation of tightness of the shoulder and lymphedema
Late radiation associated morbidity | 10 years after RT
  Incidences of fibrosis, dyspigmentation, telangiectasia, edema, arm lymph edema, range of motion of the shoulder, pain, rib fractures, pneumonitis
Patient reported outcome measures | 10 years after RT
  Rates of patient satisfaction with cosmetic outcome, body image scale, rates of depression and fear of cancer recurrence
Translational research | 10 years after RT
  Incidences of cardiac disease detected on heart CT scans, PET CT scans, and concentration of early markers of late cardiac events measured in blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Birgitte V Offersen, phd, Principal Investigator — Danish Breast cancer Cooperation Group (DBCG)
Locations (8):
- Denmark (8):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - The Danish Breast Cancer Cooperative Group, Copenhagen
  - Rigshospitalet, Copenhagen
  - Herlev Hospital, Herlev
  - Naestved Hospital, Næstved
  - Odense University Hospital, Odense
  - Vejle Hospital, Vejle

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share data when the primary and secondary endpoints have been published
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available, when the primary and secondary endpoints have been published.
Access Criteria: The research Group must apply the Danish Breast cancer Group (DBCG) to gain access to the anonymized trial data.